### **Statistical Analysis Plan**

# An Open label Study to Evaluate the Impact of Omeprazole, A Proton Pump Inhibitor, on the Pharmacokinetics of Sotorasib Coadministered with an Acidic Beverage in Healthy Volunteers

SAP Status: Final SAP Version: 1.0 SAP Date: 14 September 2022

Investigational Medicinal Product: Sotorasib (AMG 510)

Protocol Reference: 20220024

Labcorp Drug Development Study: 8493285

Sponsor: Study Site: Amgen Inc.

One Amgen Center Drive Labcorp Clinical Research Unit Inc.
Thousand Oaks, California 91320 1341 W. Mockingbird Ln., Suite 200E

Dallas, TX 75247

Information described herein is confidential and may be disclosed only with the express written permission of the sponsor.

NCT Number: NCT05497557
This NCT number has been applied to the document for purposes of posting on Clinicaltrials.gov

### TABLE OF CONTENTS

| TITLE PAGE | 1 |
|---|---|
| TABLE OF CONTENTS | 2 |
| LIST OF IN-TEXT TABLES AND FIGURES | 3 |
| LIST OF ABBREVIATIONS | 4 |
| 1. INTRODUCTION | 6 |
| 2. STUDY OBJECTIVES | 6 |
| 3. STUDY ENDPOINTS | 7 |
| 3.1. Primary Endpoints: | 7 |
| 3.2. Secondary Endpoints: | 7 |
| 4. STUDY DESIGN | 7 |
| 5. SAMPLE SIZE JUSTIFICATION | 8 |
| 6. STUDY TREATMENTS | 8 |
| 7. DEFINITIONS OF POPULATIONS | 9 |
| 7.1. All Subjects Population | 9 |
| 7.2. Safety Population | 9 |
| 7.3. Pharmacokinetic Population | 9 |
| 8. STATISTICAL METHODOLOGY | 9 |
| 8.1. General | 9 |
| 8.1.1. Handling of Data Quality Issues Due to Coronavirus Disease 2019 and Related Restrictions | |
| 8.1.2. Calculation of the Summary Statistics | 11 |
| 8.1.3. Repeat and Unscheduled Readings | 11 |
| 8.1.4. Definitions of Baseline, Change from Baseline, and Percentage Change from Baseline | 12 |
| 8.2. Subject Disposition and Population Assignment | 12 |
| 8.3. Screening Demographics | 12 |
| 8.4. Prior and Concomitant Medication | 12 |
| 8.5. Pharmacokinetic Assessments | 13 |
| 8.5.1. Pharmacokinetic Analysis | 13 |
| 8.5.2. Presentation of Pharmacokinetic Data | 15 |
| 8.5.3. Pharmacokinetic Statistical Methodology | 16 |
| 8.6. Safety and Tolerability Assessments | 16 |


Study Schematic.....8

Figure 1:


#### LIST OF ABBREVIATIONS

Abbreviations pertain to the statistical analysis plan (SAP) only (not the tables, figures, and listings [TFLs]).

ADaM Analysis Data Model

AE adverse event
ANOVA analysis of variance

AUC<sub>inf</sub> area under the plasma concentration-time curve from time zero extrapolated to

infinity

AUC<sub>0-tlast</sub> area under the plasma concentration-time curve from time zero to time of last

quantifiable concentration

BLQ below the limit of quantification

CDISC Clinical Data Interchange Standards Consortium

CI confidence interval CL/F apparent total clearance

C<sub>max</sub> maximum observed plasma concentration

COVID-19 coronavirus disease 2019 CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

CV coefficient of variation
DMP data management plan
ECG electrocardiogram

eCRF electronic case report form
GLSM geometric least squares mean

ICH International Council for/Conference on Harmonisation

LLOQ lower limit of quantification

ln natural log

LSM least squares mean

MedDRA Medical Dictionary for Regulatory Activities

PK pharmacokinetic(s)

QTcF QT interval corrected for heart rate using Fridericia's formula

SAP statistical analysis plan SD standard deviation

SDV source document verification

 $t_{1/2}$  apparent plasma terminal elimination half-life

TEAE treatment-emergent adverse event

 $\begin{array}{ll} TFL & table, figure, and listing \\ t_{lag} & absorption lag time \\ \end{array}$ 

 $t_{max}$  time of the maximum observed plasma concentration  $V_z/F$  apparent volume of distribution during the terminal phase

WHODrug World Health Organization Drug Dictionary


 $\lambda_z$  apparent terminal elimination rate constant


#### 1. INTRODUCTION

This SAP has been developed after review of the clinical study protocol (Final Protocol dated 18 May 2022) and electronic case report form (eCRF).

This SAP describes the planned analysis of the pharmacokinetic (PK), safety, and tolerability data from this study. A detailed description of the planned TFLs to be presented in the clinical study report (CSR) is provided in the accompanying TFL shells document.

In general, the analyses are based on information from the protocol, unless they have been modified by agreement with Amgen Inc. A limited amount of information about this study (eg, objectives, study design) is given to help the reader's interpretation.

This SAP must be finalized prior to the first subject enrollment (the point of enrollment occurs at the time of subject number allocation). Additionally, the SAP and TFL shells should be finalized prior to any programming activities commencing.

This SAP supersedes any statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. If additional analyses are required to supplement the planned analyses described in this SAP, they may be performed and will be identified accordingly in the CSR. Any substantial deviations from this SAP will be agreed with Amgen Inc. and identified in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E3 guideline *Structure and Content of Clinical Study Reports*, ICH E8 guideline *General Considerations for Clinical Trials*, ICH E9 guideline *Statistical Principles for Clinical Trials*, and ICH E9 R1 guideline *Addendum on Estimands and Sensitivity Analysis in Clinical Trials to the Guideline on Statistical Principles for Clinical Trials*. <sup>1,2,3,4</sup>

The document history is presented in Appendix 1.

#### 2. STUDY OBJECTIVES

The primary objective of the study is:

• to evaluate the effects of omeprazole (a PPI) and an acidic beverage on sotorasib PK when administered orally in healthy volunteers.

The secondary objective of the study is:

• to evaluate safety and tolerability of sotorasib when coadministered with omeprazole and an acidic beverage in healthy subjects.


#### 3. STUDY ENDPOINTS

#### 3.1. Primary Endpoints:

The primary endpoints of the study are sotorasib PK parameters on Days 1 and 9:

- C<sub>max</sub>
- AUC<sub>inf</sub>
- area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC<sub>last</sub>)

#### 3.2. Secondary Endpoints:

The secondary endpoints of the study are:

- adverse events
- clinical laboratory tests
- 12-lead ECGs
- vital signs.

#### 4. STUDY DESIGN

This will be a Phase 1, single-center (United States), open-label, fixed sequence study to investigate the effect of coadministration of omeprazole with an acidic beverage on the PK of sotorasib in healthy male and healthy female subjects. Up to 14 subjects will be enrolled to ensure that 12 subjects complete the study. All subjects will receive each of the following treatments:

- Day 1: 960 mg sotorasib (8 x 120 mg tablets) administered orally with 240 mL of water after an overnight fast of at least 10 hours
- Days 4 to 8: 40 mg omeprazole (delayed release capsule) administered orally with 240 mL of water QD after an overnight fast of at least 10 hours
- Day 9: 40 mg omeprazole (delayed release capsule) followed by 960 mg sotorasib (8 x 120 mg tablets) administered orally within 5 minutes with 240 mL of an acidic beverage after an overnight fast of at least 10 hours.


**CONFIDENTIAL** Protocol Reference: 20220024

An overview of the study design is shown in Figure 1.

Figure 1: **Study Schematic** 



Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. Subjects will be admitted into the Clinical Research Unit (CRU) on Day -1 and be confined to the CRU until discharge/end of study (EOS) on Day 11.

The total duration of study participation for each subject (from Screening through EOS visit) is anticipated to be approximately 5.5 weeks.

The start of the study is defined as the date the first enrolled subject signs an Informed Consent Form (ICF). The point of enrollment occurs at the time of subject number allocation. The end of the study is defined as the date of the last subject's last assessment (scheduled or unscheduled).

#### 5. SAMPLE SIZE JUSTIFICATION

Approximately 14 subjects will be enrolled in order that approximately 12 subjects complete the study. The sample size for this study was based upon precedent set by other PK studies of a similar nature and was not based on power calculations.

#### 6. STUDY TREATMENTS

The study treatment names, abbreviations, and ordering to be used in the TFLs are presented in Table 1.

**Table 1: Presentation of Study Treatments in TFLs** 

| Study Treatment | Order in TFLs |
|---|---|
| Sotorasib administered alone | 1 |
| Omeprazole coadministered with Sotorasib and an acidic beverage | 2 |

All TFLs will be based on actual treatments (eg, if subject was assigned to receive placebo but was wrongfully dosed with active treatment they would be summarized and listed under active treatment).

#### 7. DEFINITIONS OF POPULATIONS

Any protocol deviations, including those due to coronavirus disease 2019 (COVID-19) and related restrictions (see Section 8.1.1), will be considered prior to database lock for their importance and taken into consideration when assigning subjects to populations.

#### 7.1. All Subjects Population

The all subjects population will include all subjects who signed the ICF and had any study assessment recorded in the database per the protocol.

#### 7.2. Safety Population

The safety population will include all subjects who received at least 1 dose of sotorasib and have at least 1 postdose safety assessment.

#### 7.3. Pharmacokinetic Population

The PK population will include all subjects who received at least 1 dose of sotorasib and have evaluable PK data. The PK population for the primary endpoint analysis will include all subjects who received both sotorasib, and sotorasib in combination with omeprazole and an acidic beverage, and have evaluable PK data. A subject will be excluded from the PK summary statistics and statistical analysis if the subject has an adverse event of vomiting that occurs at or before 2 times median t<sub>max</sub> or diarrhea within 24 hours of dosing.

#### 8. STATISTICAL METHODOLOGY

#### 8.1. General

Listings will be provided for all data captured in the database, with the exception of medical history. Listings will include all subjects assigned to the all subjects population and include data up to the point of study completion or discontinuation. Subjects are generally considered to have completed the study if they complete the scheduled follow-up visit (rather than early termination visit). Any subject who discontinues the study will be identified accordingly in the listings. Summaries and statistical analyses will include the subjects assigned to the relevant population based on data type.


Data analysis will be performed using the SAS® statistical software package Version 9.4 (or higher if a new version is issued during the study).

Analysis Data Model (ADaM) datasets will be prepared using Clinical Data Interchange Standards Consortium (CDISC) ADaM Version 2.1 (or higher if a new version is issued during the study) and CDISC ADaM Implementation Guide Version 1.1 (or higher if a new version is issued during the study). Pinnacle 21 Community Validator Version 4.0.1 (or higher if a new version is issued during the study) will be utilized to ensure compliance with CDISC standards.

For all statistical analyses, the hypothesis testing will be two one-sided t-test with each side tested on 0.05 significance level, unless specifically stated otherwise.

Where reference is made to 'valid' data, this refers to non-missing data which meet the predetermined criteria (eg, are not flagged for exclusion).

Where reference is made to 'all calculations', this includes, but is not limited to, summary statistics, statistical analyses, baseline derivation, changes from baseline and percentage changes from baseline.

All figures will be produced on linear-linear or discrete-linear scales, as applicable, unless specifically stated otherwise.

### 8.1.1. Handling of Data Quality Issues Due to Coronavirus Disease 2019 and Related Restrictions

Due to COVID-19 and related restrictions, there is a high risk for impact to data integrity, with the recognized potential for:

- Missed visits, caused by, for example:
  - Subject unable to travel to site due to restrictions, the need to quarantine, or COVID-19 infection
  - o Subject unwilling to go to site due to fear of COVID-19 infection
  - o Site postponing subject's visit due to investigator not being available (eg, if they have been dispatched to hospital handling COVID19 infections)
- Site unable to replenish supply of investigational product
- Incomplete data entry by sites due to limited resources to support study or no access to source documents or to eCRF
- Outstanding source document verification (SDV) due to sponsor or country restrictions on remote SDV, or no or limited access to site(s) for on-site visits
- Unanswered queries


At the time of the reporting of the study results, all protocol deviations due to COVID-19 or related restriction will be assessed for their severity and impact on the analyses. If needed, appropriate statistical methods will be applied as a mitigating action (eg, data might be categorized into 2 analysis groups, with and without COVID-19 and related restrictions impact); however, this will exclude any imputations of the missing values. Any mitigating actions will be agreed with Amgen Inc in advance and identified in the CSR.

#### 8.1.2. Calculation of the Summary Statistics

For continuous data the following rules will be applied:

- Missing values will not be imputed, unless specifically stated otherwise.
- Unrounded data will be used in the calculation of summary statistics.
- If the number of subjects with valid observations (n) <3, summary statistics will not be calculated, with the exception of n, minimum, and maximum.
- In general, as early termination data are not associated with any scheduled timepoint, they will be excluded from all calculations of summary statistics and statistical analyses. Exceptions may be made where justified.

For categorical data the following rules will be applied:

- For ordered categorical data (eg, adverse event [AE] severity), all categories between the possible minimum and maximum categories will be included, even if n = 0 for a given category.
- For non-ordered categorical data (eg, race), only those categories for which there is at least 1 subject represented will be included; unless specifically stated otherwise.
- Missing values will not be imputed, unless specifically stated otherwise. A 'missing' category will be included for any parameter for which information is missing. This will ensure that the population size totals are consistent across different parameters.

#### 8.1.3. Repeat and Unscheduled Readings

For vital signs and 12-lead ECG data only, any predose value recorded in addition to the original value or a postdose value recorded within 15 minutes of the original value will be defined as a repeat value; any postdose value recorded more than 15 minutes after the original value will be defined as an unscheduled value. For all other data types (eg, laboratory parameters), any value recorded in addition to the original value will be defined as an unscheduled value.

The original value will be replaced by the last associated repeat value in all calculations.


As unscheduled values are not associated with any scheduled timepoint, they will be excluded from all calculations, with the exception of the baseline derivation (see

Section 8.1.4) and 12-lead ECG outlier analysis (see Section 8.6.4).

# 8.1.4. Definitions of Baseline, Change from Baseline, and Percentage Change from Baseline

The baseline will be defined as the last value recorded prior to dosing. If the date/time of the value is incomplete or missing, it will be excluded from the baseline calculation, unless the incomplete date/time indicates the value was recorded prior to dosing.

Individual changes from baseline will be calculated by subtracting the individual subject's baseline value from the value at the postdose timepoint.

Individual percentage changes from baseline will be calculated by subtracting the individual subject's baseline value from the value at the postdose timepoint, then dividing this calculated value by the individual subject's baseline value and multiplying by 100.

The summary statistics for change from baseline and percentage changes from baseline will be derived from individual subjects' values (eg, mean change from baseline will be the mean of the individual changes from baseline for all subjects, rather than difference between the mean value at the postdose timepoint and mean value at baseline).

See Section 8.1.3 for more detail on handling repeat and unscheduled readings in the calculations.

#### 8.2. Subject Disposition and Population Assignment

Subject disposition and population assignment will be listed.

A summary table by treatment will be provided, based on the safety population.

#### 8.3. Screening Demographics

The screening demographics including age, sex, race, ethnicity, height, body weight, and body mass index will be listed.

A summary table by treatment will be provided, based on the safety population.

#### 8.4. Prior and Concomitant Medication

Prior medication will be defined as medication that ends prior to the first dose. Concomitant medication will be defined as medication that starts during or after the first dose or starts but does not end prior to the first dose.

Prior and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHODrug) Global, Format B3, Version March 2022 (or later if a new version is


issued during the study; see the data management plan [DMP] for more details). Prior and concomitant medications will be listed.

#### 8.5. Pharmacokinetic Assessments

#### 8.5.1. Pharmacokinetic Analysis

The following PK parameters will be determined where possible from the plasma concentrations of sotorasib using noncompartmental methods in validated software program Phoenix WinNonlin (Certara, Version 8.1.1 or higher):

| Parameter | Unitsa | Definition |
|---|---|---|
| AUC <sub>0-tlast</sub> | h*ng/mL | area under the concentration-time curve from time 0 to the time of the last quantifiable concentration $(t_{last})^b$ |
| $AUC_{inf}$ | h*ng/mL | area under the concentration-time curve from time 0 extrapolated to infinity <sup>c</sup> |
| $C_{\text{max}}$ | ng/mL | maximum observed concentration |
| $t_{max}$ | h | time of the maximum observed concentration |
| $t_{last}$ | h | time of the last quantifiable concentration |
| $t_{1/2}$ | h | apparent terminal elimination half-life |
| CL/F | L/h | apparent total clearance |
| $V_z/F$ | L | apparent volume of distribution during the terminal phase |

<sup>&</sup>lt;sup>a</sup> Units are based on concentration units (provided by the bioanalytical lab or preferred units for presentation of PK parameters) and dose units used in the study.

Additional PK parameters may be determined where appropriate.

Pharmacokinetic analysis will be carried out where possible using actual blood sampling times postdose. If an actual time is missing, the sample concentration result will be treated as missing unless there is scientific justification to include the result using the nominal time.

The parameters  $C_{max}$ ,  $t_{last}$ , and  $t_{max}$  will be obtained directly from the concentration-time profiles. If  $C_{max}$  occurs at more than 1 timepoint,  $t_{max}$  will be assigned to the first occurrence of  $C_{max}$ .

# 8.5.1.1. Criteria for the Calculation of Apparent Terminal Elimination Rate Constant and Half-life

The start of the terminal elimination phase for each subject will be defined by visual inspection and generally will be the first point at which there is no systematic deviation from the log-linear decline in concentrations.

The apparent terminal elimination rate constant  $(\lambda_z)$  will only be calculated when a reliable estimate can be obtained using at least 3 data points, preferably not including  $C_{max}$ , and the adjusted coefficient for determination of exponential fit (R<sup>2</sup>-adj) of the regression line is  $\geq 0.8$ .


<sup>&</sup>lt;sup>b</sup> The AUC will be calculated using the linear trapezoidal (linear interpolation) rule.

<sup>&</sup>lt;sup>c</sup> Based on the last observed quantifiable concentration

calculated if the  $R^2$ -adj value of the regression line is >0.8.

Labcorp Drug Development Study: 8493285 Protocol Reference: 20220024 Parameters requiring  $\lambda_z$  for their calculation (eg, AUC<sub>0-\infty</sub>, t<sub>1/2</sub>, CL/F, V<sub>z</sub>/F) will only be

The following regression-related diagnostic PK parameters will be determined, when possible:

| Parameter | Units | Definition |
|---|---|---|
| %AUC <sub>extrap</sub> | % | percentage of AUC due to extrapolation from the last quantifiable concentration to infinity |
| $\lambda_z$ | 1/h | apparent terminal elimination rate constant |
| $\lambda_z$ Upper | h | end of exponential fit |
| $\lambda_z$ Lower | h | start of exponential fit |
| $\lambda_z N$ | NA | number of data points included in the log-linear regression |
| $\lambda_z$ Span Ratio | NA | time period over which $\lambda_z$ was determined as a ratio of $t_{\mbox{\scriptsize 1/2}}$ |
| R <sup>2</sup> -adj | NA | adjusted coefficient for determination of exponential fit |

Where possible, the span of time used in the determination of  $\lambda_z$  (ie, the difference between  $\lambda_z$  Upper and  $\lambda_z$  Lower) should be  $\geq 2$  half-lives. If the  $\lambda_z$  Span Ratio is  $\leq 2$ , the robustness of the  $t_{1/2}$  values will be discussed in the clinical study report (CSR).

# 8.5.1.2. Criteria for Calculation and Reporting of Area Under the Concentration-time Curve

The minimum requirement for the calculation of area under the concentration-time curve (AUC) will be the inclusion of at least 3 consecutive concentrations above the lower limit of quantification. If there are only 3 consecutive concentrations, at least 1 should follow  $C_{\text{max}}$ . An exception may be made for metabolites, where  $C_{\text{max}}$  may be the last timepoint.

If the extrapolated area is >20%, AUC<sub>inf</sub> (and derived parameters) will be listed but flagged and excluded from statistics.

If AUC<sub>inf</sub> cannot be determined reliably for all subjects, an alternative AUC measure, such as AUC to a fixed timepoint or AUC<sub>0-tlast</sub>, may be used in the statistical analysis.

# 8.5.1.3. Criteria for Handling Concentration Below the Limit of Quantification or Missing Concentrations for Pharmacokinetic Analysis

Plasma concentrations below the limit of quantification (BLQ) will be assigned a value of 0 before the first measurable concentration and thereafter BLQ concentrations will be treated as missing. The following rules apply to the specific situations defined below:

- If an entire concentration-time profile is BLQ, it will be excluded from PK analysis.
- Where 2 or more consecutive concentrations are BLQ at the end of a profile, the profile will be deemed to have terminated and any further quantifiable concentrations will be


set to missing for the calculation of the PK parameters, unless they are considered to be a true characteristic of the profile of the drug.

• If a predose plasma concentration is missing, it will be set to 0 by default within Phoenix WinNonlin.

#### 8.5.1.4. Treatment of Outliers in Pharmacokinetic Analysis

If a value is considered to be anomalous due to being inconsistent with the expected PK profile, it may be appropriate to exclude the value from the PK analysis. However, the exclusion of any data must have strong justification and will be documented in the CSR.

Any quantifiable predose concentration value in the first treatment period will be considered anomalous and set to missing for the PK analysis. This will be set to 0 by default in Phoenix WinNonlin.

If the predose concentration is >5% of  $C_{max}$  in the second treatment period, all PK concentration and parameter data will be excluded from the summary statistics and statistical analysis for that period.

#### 8.5.2. Presentation of Pharmacokinetic Data

All PK concentrations and parameters will be listed.

Summary tables, arithmetic mean (+ standard deviation [SD]) figures, overlaying individual figures, and individual figures by treatment and time postdose will be provided for plasma PK concentrations. All figures will be produced on both linear-linear and linear-logarithmic scales, with the exception of figures across all days, which will be produced on the linear-linear scale only. The +SD bars will only be displayed on the linear-linear scale.

Summary tables by treatment will be provided for all PK parameters, with the exception of diagnostic regression-related PK parameters. Separate summary tables by treatment and time interval will be provided for excretion parameters and cumulative excretion parameters.

A subject may be excluded from the PK summary statistics and statistical analysis if the subject has an AE of vomiting that occurs at or before 2 times the median  $t_{max}$ .

If the actual time of sample collection deviates from the nominal time by more than  $\pm 10\%$ , the concentration will be flagged, but included in the summary statistics.

Individual concentrations deemed to be anomalous will be flagged in the listings and excluded from the summary statistics.

For plasma concentration data the following rules will apply:

- Values that are BLQ will be set to 0 for the calculation of summary statistics.
- Arithmetic mean or median values that are BLQ will be presented as 0.


For PK parameters the following rule will apply:

• Geometric mean and coefficient of variation will not be calculated for t<sub>last</sub>, t<sub>max</sub>.

#### 8.5.3. Pharmacokinetic Statistical Methodology

A statistical analysis will be conducted to investigate the drug-drug interaction, the primary PK parameters will be AUC<sub>inf</sub>, AUC<sub>0-tlast</sub>, and C<sub>max</sub> for sotorasib on each of the dosing days. All other PK parameters will be regarded as secondary and will not be subject to inferential statistical analysis.

A linear mixed effects model will be used to analyze log-transformed primary PK parameters. The model will assume fixed effect for treatment and a random effect for subject. Geometric mean ratios for  $C_{max}$  and AUC values and associated 90% confidence intervals (Test/Reference) will be estimated. The "Reference" treatment for PK analysis will be sotorasib administered alone with water, while the "Test" treatment will be omeprazole administered in combination with sotorasib and an acidic beverage.

For each PK parameter separately, the least squares mean (LSM) for each treatment, difference in LSMs between the test and reference treatments, and corresponding 90% confidence interval (CI) will be calculated; these values will then be back-transformed to give the geometric least squares mean (GLSM), ratio of GLSMs, and corresponding 90% CI.

Additionally, the pooled estimate (across all treatments) of the within-subject CV will be calculated, and residual plots will be produced to assess the adequacy of the model(s) fitted.

Examples of the SAS code that will be used are as follows:

#### **Mixed Model Analysis**

```
proc mixed data = <data in>;
  by parcatln parcatl pkday paramn param;
  class trtan usubjid;
  model l_pk = trtan aperiod trtseqp / cl residual ddfm = kr;
  lsmeans trtan / cl pdiff = control('1') alpha = 0.1;
  random intercept / subject = usubjid(trtseqp);
  ods output lsmeans = <data out>;
  ods output diffs = <data out>;
  ods output covparms = <data out>;
run;
```

#### 8.6. Safety and Tolerability Assessments

#### 8.6.1. Adverse Events

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 25.0. (or higher if a new version is issued during the study; see the DMP for more details).

A treatment-emergent adverse event (TEAE) will be defined as an AE that starts during or after the first dose, or starts prior to the first dose and increases in severity after the first dose.


A treatment related TEAE will be defined as a TEAE with a relationship of possibly related or related to the study treatment, as determined by the investigator.

All AEs will be listed. In addition to the data recorded in the database, the listings will include derived onset time and duration. Onset time will be calculated from the time of dosing for TEAEs only.

The frequency of subjects with TEAEs and the number of TEAEs will be summarized for the following categories:

- TEAEs (overall, serious, leading to discontinuation, and leading to death) by treatment
- TEAEs by severity and treatment
- Treatment-related TEAEs (overall, serious, leading to discontinuation, and leading to death) by treatment
- Treatment-related TEAEs by severity and treatment

The frequency of subjects will be summarized separately for TEAEs and treatment-related TEAEs by the following:

- System organ class, preferred term, severity and treatment
- Preferred term, severity and treatment

For the AE data the following rules will apply:

- For the derivation of TEAE status: If the start date/time of an AE is incomplete or missing, an AE will be assumed to be a TEAE, unless the incomplete start date/time or the end date/time indicates an AE started prior to the first dose.
- For the derivation of treatment-related TEAE status: If the study treatment relationship for a TEAE is missing, a TEAE will be assumed to be a treatment-related TEAE.
- For the derivation of onset time (applicable to TEAEs only): If the start date/time of a TEAE is missing, onset time will not be calculated. If the start date/time of a TEAE is incomplete, where possible, the minimum possible onset time will be calculated and presented in '≥DD:HH:MM' format (eg, if the date/time of the last associated dose is 01MAY2019/08:00 and recorded start date/time of a TEAE is 03MAY2019, then the minimum possible onset time will be calculated by assuming a TEAE started at the first hour and minute of 03MAY2019 [03MAY2019/00:00], thus will be presented as onset time ≥01:16:00 in the listing). If the start date of a TEAE is the same as the date of the last associated dose but the start time of a TEAE is missing, an onset time will be presented as '≥00:00:01'. Any clock changes will be accounted for in the derivation.
- For the derivation of duration (applicable to all AEs): If the end date/time of an AE is missing, duration will not be calculated. If the start or end date/time of an AE is


Protocol Reference: 20220024


incomplete, where possible, the maximum possible duration will be calculated and presented in '\(\leq\)DD:HH:MM' format (eg, if the start of an AE date/time is 01MAY2019/08:00 and its recorded end date/time is 03MAY2019, then the maximum possible duration will be calculated by assuming an AE ended at the last hour and minute of 03MAY2019 [03MAY2019/23:59], thus will be presented as duration \(\leq\)02:15:59 in the listing). Any clock changes will be accounted for in the derivation.

- For the calculation of TEAE summary statistics: If the severity of a TEAE is missing, that TEAE will be counted under the 'missing' category.
- For the calculation of TEAE summary statistics: If a subject experienced multiple TEAEs with the same preferred term for the same treatment, this will be counted as 1 TEAE for that treatment under the maximum severity recorded.

#### 8.6.2. Clinical Laboratory Parameters

All clinical laboratory parameters, their changes from baseline, and percentage changes from baseline will be listed, as applicable; any value outside the clinical reference range will be flagged. Separate listings will be provided for any parameter for which there is any individual subject value outside the respective clinical reference range.

Summary tables by timepoint will be provided for clinical chemistry, hematology, and urinalysis parameters, with changes from baseline and percentage changes from baseline, as applicable.

Values recorded as  $\langle x, \leq x, \rangle x$ , or  $\geq x$  will be displayed in the listings as recorded. For the derivation of listing flags and calculation of summary statistics,  $\langle x \rangle x$  and  $\leq x \rangle x$  values will be set to 0, whereas  $\geq x$  and  $\geq x \rangle x$  values will be set to x.

#### 8.6.3. Vital Signs Parameters

All vital signs parameters, their changes from baseline, and percentage changes from baseline, will be listed, as applicable; any value outside the clinical reference range will be flagged.

Summary tables by timepoint will be provided for all vital signs parameters, with changes from baseline and percentage changes from baseline, as applicable.

#### 8.6.4. 12-lead Electrocardiogram Parameters

All 12-lead ECG parameters will be listed, as applicable; any value outside the clinical reference range will be flagged.

Summary tables by timepoint will be provided for all 12-lead ECG parameters.


Protocol Reference: 20220024


An outlier analysis will be performed for QT interval corrected for heart rate using Fridericia's formula (QTcF). The analysis will include all individual original, repeat, and unscheduled postdose values.

The maximum postdose values will be summarized by treatment according to the following categories:

- ≤450 ms
- >450 and ≤480 ms (all instances flagged in the listing)
- >480 and ≤500 ms (all instances flagged in the listing)
- >500 ms (all instances flagged in the listing)

The maximum increases from baseline will be summarized by treatment according to the following categories:

- ≤30 ms
- >30 and  $\le 60$  ms (all instances flagged in the listing)
- >60 ms (all instances flagged in the listing)

#### 8.6.5. Other Assessments

Medical history will not be listed.

All other safety and tolerability assessments not detailed in the above sections will be listed only.

#### 8.6.6. Safety and Tolerability Statistical Methodology

No inferential statistical analyses are planned.

#### 9. INTERIM ANALYSES

No formal interim analyses are planned for this study.

#### 10. SIGNIFICANT CHANGES FROM THE PROTOCOL-SPECIFIED ANALYSES

There were no significant changes from the protocol-specified analyses.

#### 11. REFERENCES

1. ICH. ICH Harmonised Tripartite Guideline: Structure and content of clinical study reports (E3). 30 November 1995.


17 July 1997.

- Protocol Reference: 20220024 2. ICH. ICH Harmonised Tripartite Guideline: General considerations for clinical trials (E8).
- 3. ICH. ICH Harmonised Tripartite Guideline: Statistical principles for clinical trials (E9). 5 February 1998.
- 4. ICH. ICH Harmonised Tripartite Guideline: Addendum on estimands and sensitivity analysis in clinical trials to the guideline on statistical principles for clinical trials (E9 [R1]). 20 November 2019


#### 12. APPENDICES

### **Appendix 1: Document History**

| Status and Version Date of Change | | Summary/Reason for Changes |
|-----------------------------------|----|----------------------------|
| Final Version 1.0 | NA | NA; the first version. |

NA = not applicable


# Statistical Analysis Plan (SAP)/Initiation of Programming Approval Form

| Sponsor Name: | Amgen Inc. | | |
|---|---|---|---|
| Sponsor Protocol/CIP II | 2 1220024 | Covanc<br>e Study<br>ID: | 8493285 |
| SAP text filename: | AMG<br>510_20220024_8493285<br>_SAP_Final_14sept2022 | TFL<br>shells<br>filenam<br>e: | AMG<br>510_20220024_8493285<br>TFL<br>shells_final_14sept2022 |
| Version: | 1 | Date: | 9/20/2022 |
| Approval Signature | | | |
| Print Name<br>Job Title | | | |
| Date | | | |
| C | | | |
| signatories agree to the the associated tables, programming of the Andocuments can proceed signing may result in a signing may result in a significant signature. Approval Signature Print Name Job Title | n the statistical analysis place analyses to be performed figures, and listings (TFLs) allysis Dataset Model (ADaM) d. Any modifications to the Solwork-scope change. | for this sto<br>Once the<br>datasets | udy and to the format o<br>e SAP has been signed,<br>and TFLs based on these |
| By signing below whe signatories agree to the the associated tables, programming of the Andocuments can proceed signing may result in a Approval Signature Print Name | e analyses to be performed in figures, and listings (TFLs) alysis Dataset Model (ADaM) d. Any modifications to the Solution work-scope change. | for this sto<br>Once the<br>datasets | udy and to the format of<br>e SAP has been signed,<br>and TFLs based on these |
| By signing below whe signatories agree to the the associated tables, programming of the Andocuments can proceed signing may result in a signing may result in a significant of the Approval Signature Print Name Job Title Date | e analyses to be performed in figures, and listings (TFLs) alysis Dataset Model (ADaM) d. Any modifications to the Solution work-scope change. | for this sto<br>Once the<br>datasets<br>SAP text and | udy and to the format of<br>e SAP has been signed,<br>and TFLs based on these<br>nd TFL shells made after |
| By signing below whe signatories agree to the the associated tables, programming of the Andocuments can proceed signing may result in a signing may result in a significant of the Approval Signature Print Name Job Title Date | e analyses to be performed if figures, and listings (TFLs) alysis Dataset Model (ADaM) d. Any modifications to the Solwork-scope change. | for this sto<br>Once the<br>datasets<br>SAP text and | udy and to the format of<br>e SAP has been signed,<br>and TFLs based on these<br>nd TFL shells made after |

### 16.1.9.2. Quality Tolerance Limit Definitions

| Parameter | Justification for Parameter | Unit Tolerance |
|---|---|---|
| Minimum number of evaluable subjects needed. | A shortfall in the overall number of subjects could have had a significant impact on interpretation of the primary endpoint because of limited/insufficient exposure. | N: 14 |


Protocol Reference: 20220024

Final 